CLINICAL TRIAL: NCT02564016
Title: Efficacy of Labor Epidurals for Postpartum Tubal Ligation: Effect of Postpartum Epidural Saline Infusion on the Reactivation of Labor Epidurals for Postpartum Tubal Ligation Following Vaginal Delivery
Brief Title: Efficacy of Labor Epidurals for Postpartum Tubal Ligation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Of 36 participants only 8 participants able to fully complete the study procedures. At this time, the study will be closed due to poor enrollment numbers.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033454
Record Dates: First submitted 2015-07-17; First posted 2015-09-30 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capped Epidural (Active Comparator): Group 1 (control) will have the epidural catheter capped and left in place.
  Interventions: Other: Capped Epidural
- Normal Saline Infusion (Experimental): Group 2 (treatment) will have an epidural infusion initiated with preservative-free normal saline at a continuous rate of 4ml/hour
  Interventions: Drug: Normal Saline Infusion

INTERVENTIONS:
Drug: Normal Saline Infusion — Group 2 (treatment) will have an epidural infusion initiated with preservative-free normal saline at a continuous rate of 4ml/hour
  Other Names: 0.9% Sodium Chloride
  Arms: Normal Saline Infusion
Other: Capped Epidural — epidural will be capped with no saline infusion.
  Arms: Capped Epidural

SUMMARY:
The goal of this study is to evaluate the effect of continuous postpartum epidural saline infusion on the reactivation of labor epidurals for postpartum tubal ligation surgery following vaginal delivery.

DETAILED DESCRIPTION:
The aim of this research is to determine the effect of postpartum epidural saline infusion on the reactivation of labor epidural catheters which are used as the anesthetic technique for PPTL following vaginal delivery. It is proposed that continuous epidural saline infusion will decrease the incidence of catheter obstruction by preventing clot, fibrosis, or tissue plugging and therefore improve reactivation rates. To our knowledge, this is a novel method for attempting to improve epidural reactivation rate and if successful, it would challenge the current practice of only capping epidurals following delivery and later attempting reactivation prior to PPTL. This may, possibly, become a new technique used to improve the rate of epidural reactivation for PPTL.

If study results show improved labor epidural reactivation rates, benefits would include decreased patient morbidity and greater patient comfort and satisfaction by avoiding the risks of additional neuraxial procedures as well as general anesthesia. These risks include difficult or failed intubation, aspiration, hypotension, headache, postoperative nausea and vomiting, and sore throat. Improving epidural reactivation rate could also result in greater OR efficiency and decreased costs for the patient and hospital.

The investigators also hope to elucidate factors associated with catheter migration or dislodgement and subsequent failure of epidural reactivation. Additionally, we hope to determine what effect obesity and length of time prior epidural reactivation have on epidural reactivation rates.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18 to 45 years of age
* Admitted to MUSC in labor or for induction of labor resulting in a vaginal delivery epidural analgesia
* Postpartum tubal ligation following delivery
* American Society of Anesthesiologists (ASA) Physical Class 1, 2, and 3

Exclusion Criteria:

* Critically Ill Patients (patients admitted to the ICU)
* Cognitively Impaired Persons (patients with a diagnosis of cognitive deficit)
* Cesarean delivery
* Punctured dura
* Patients enrolled in other epidural research studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Roberts, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capped Epidural | Normal Saline Infusion
Started | 22 | 14
Completed | 4 | 4
Not Completed | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capped Epidural | Normal Saline Infusion | Total
Number analyzed (Participants) | 22 | 14 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 14 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [21 to 42] | 32 [22 to 41] | 32 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 14 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Epidural Reactivation
Description: The goal of this study is to evaluate the effect of continuous postpartum epidural saline infusion on the reactivation of labor epidurals for postpartum tubal ligation surgery following vaginal delivery.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Capped Epidural | Normal Saline Infusion
Number analyzed (Participants) | 22 | 14
participants | 3 | 4

2. Secondary Outcome: Count of Participants Whose BMI Affected the Reactivation Rate of Labor Epidurals for Postpartum Tubal Ligation Surgery Following Vaginal Delivery.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Capped Epidural | Normal Saline Infusion
Number analyzed (Participants) | 22 | 14
Participants | 4 | 4

3. Secondary Outcome: Count of Participants Who Experienced Epidural Reactivation Failure
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Capped Epidural | Normal Saline Infusion
Number analyzed (Participants) | 22 | 14
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: The timeframe is approximately 1-4 days.
Arm/Group | Capped Epidural | Normal Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/14
Other Adverse Events (participants affected / at risk) | 0/22 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No